CLINICAL TRIAL: NCT03059771
Title: Mobile Enhancement of Motivation in Schizophrenia: A Pilot Trial of a Personalized Text Message Intervention for Motivation Deficits
Brief Title: Mobile Enhancement of Motivation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other); American Psychological Foundation (Other); Indiana University-Purdue University Indianapolis Department of Psychology (Unknown)
Responsible Party: Principal Investigator, Michelle Salyers, Professor and Director of Clinical Psychology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1701070796
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Micro-Electrical-Mechanical Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Enhancement of Motivation (MEMS) (Experimental): Facilitators will first collaboratively help participants set personal recovery-goals using Collaborative Goal Technology (Clarke et al., 2006). Participants will then receive three sets of interactive text messages each weekday for eight weeks to reinforce and cue goal completion.
  Interventions: Behavioral: Mobile Enhancement of Motivation (MEMS)
- Control (Active Comparator): Participants will only engage in a goal-setting session where facilitators will collaboratively help participants set personal recovery-goals using Collaborative Goal Technology (Clarke et al., 2006).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Mobile Enhancement of Motivation (MEMS) — The MEMS group will engage in a goal-setting session and then receive personalized text-messages to support goal attainment.
  Arms: Mobile Enhancement of Motivation (MEMS)
Behavioral: Control — The control group will only engage in a goal-setting session.
  Arms: Control

SUMMARY:
Motivation deficits are a strong determinant of poor functional outcomes in people with schizophrenia. Mobile interventions are a promising approach to improving these deficits, as they can provide frequent cues and reinforcements that support goal-directed behavior. The primary aims of this study are to conduct a pilot study using a randomized design to 1) Test the feasibility and acceptability of a personalized mobile text message intervention, Mobile Enhancement of Motivation in Schizophrenia (MEMS) and to 2) Test the preliminary effectiveness of MEMS compared to a control condition.

DETAILED DESCRIPTION:
Objectives: Motivation deficits are one of the strongest determinants of poor functional outcomes in people with schizophrenia. Mobile interventions are a promising approach to improving these deficits, as they can provide frequent cues and reinforcements that support goal-directed behavior. The objective of this study is to conduct a pilot study using a randomized design to 1) Test the feasibility and acceptability of a personalized mobile text message intervention, Mobile Enhancement of Motivation in Schizophrenia (MEMS) and to 2) Test the preliminary effectiveness of MEMS compared to a control condition. Methods: Up to forty outpatients with a schizophrenia-spectrum disorder will be recruited. All participants will set individualized recovery goals to complete over an eight-week period; those randomized to receive MEMS will also receive three sets of personalized, interactive text messages each weekday to reinforce and cue goal completion. Before and after the eight-week period, participants in both groups will complete validated measures of motivation. Both groups will also report their goal attainment after eight weeks. Results: It is anticipated that those in the MEMS group will demonstrate greater goal attainment and improvements in motivation compared to the control group. Discussion: This project will test the initial feasibility, acceptability, and effectiveness of a novel intervention for improving one of the most debilitating aspects of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia-spectrum diagnosis
* Have a text-message enabled cell-phone
* Are a current client at a participating community mental health center
* Are in a non-acute phase of illness or have no medication changes or hospitalizations in the prior 30 days
* Demonstrate a minimum of moderate motivation impairments according to the Clinical Assessment Interview for Negative Symptoms (CAINS; Kring et al., 2013)
* Have an English reading level at or above the fourth grade according to the Graded Word List (Pray & Ross, 1969)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Goal completion | follow-up (8 weeks)
  The percentage of baseline goals participants completed over the eight-week period will be assessed at the follow-up assessment.

SECONDARY OUTCOMES:
Motivation and Pleasure Scale-Self-Report (MAP-SR) | baseline and follow-up (8 weeks)
  The MAP-SR is a self-report measure 15-item self-report measure that assesses participant's level of motivation and pleasure in several domains, including work and recreational activities. It has been found to be valid and reliable in a schizophrenia-spectrum sample (Llerena, et al., 2013).
Intrinsic Motivation Index | baseline and follow-up (8 weeks)
  The 3-item Intrinsic Motivation Index (Nakagami et al., 2008) from the clinician-rated Quality of Life Scale (Heinrichs et al., 1984) will be used to assess trait-like intrinsic motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Midtown Community Mental Health Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Luther L, Fischer MW, Johnson-Kwochka AV, Minor KS, Holden R, Lapish CL, McCormick B, Salyers MP. Mobile enhancement of motivation in schizophrenia: A pilot randomized controlled trial of a personalized text message intervention for motivation deficits. J Consult Clin Psychol. 2020 Oct;88(10):923-936. doi: 10.1037/ccp0000599. Epub 2020 Aug 13. PMID 32790451